CLINICAL TRIAL: NCT03474783
Title: To Explore the Factors Affecting the Effectiveness of Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathay General Hospital (Other)
Responsible Party: Principal Investigator, Cathay General Hosp. IRB, Nursing Supervisor, Cathay General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CGH-P 104061
Record Dates: First submitted 2018-03-15; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multidisciplinary intervention (Experimental)
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Stages of change of intentions to cease smoking of participants at the baseline were determined, and a personal-tailored health education was accordingly delivered.

SUMMARY:
Objectives:

Promoting quitting smoking and training smoking cessation educators in hospital, school, community, and workplace was being vigorously pushed by Health Promotion Administration. Since the implementation of the second-generation smoking cessation program by Health Promotion Administration, both the general public and medical institutions have worked with greater vitality to practice and promote quitting smoking. However, studies on smoking cessation in the inpatient remain inadequate. Increasing cessation motivation for inpatient smokers and evaluating their nicotine dependence are essential. In this study, we aimed to explore the factors that might influence the smoking cessation in the inpatients.

Method: A cross-sectional questionnaire survey was conducted on inpatients participants at the smoking cessation.

Questionnaire comprising（1）Demographic characteristics: age, sex, marital status, education, （2）physiological factors（concentration of carbon monoxide, nicotine dependence, disease severity）,（3）psychological factors（psychological dependence on smoking , smoking cessation stages of behavior change, smoking cessation self-efficacy）, （4）Social Factor: social support,（5）smoking Behavior indicators: smoked, daily cigarette consumption, smoking experience. After giving health education cessation of treatment one month, three months and six months, interviewed by telephone quitting behavior index contains daily cigarette consumption, quit rates point.

ELIGIBILITY:
Inclusion Criteria:

* being a current smoker (who had smoked more than 100 cigarettes in their lifetime),
* aged > 20 years,
* with clear consciousness,
* being able to communicate using Mandarin or Taiwanese

Exclusion Criteria:

* with acute psychiatric disorders,
* inability to complete the questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
point prevalence abstinence | 1 month after intervention
  whether quitting smoking

SECONDARY OUTCOMES:
point prevalence abstinence | 3 months after intervention
  whether quitting smoking
point prevalence abstinence | 6 months after intervention
  whether quitting smoking

IPD SHARING:
Plan to Share IPD: No